CLINICAL TRIAL: NCT00747604
Title: Increlex® (Mecasermin [rDNA Origin] Injection) Growth Forum Database - IGFD Registry: A Patient Registry for Monitoring Long-term Safety and Efficacy of Increlex
Brief Title: IGFD Registry: A Patient Registry for Monitoring Long-term Safety and Efficacy of Increlex
Status: Terminated | Type: Observational
Why Stopped: Shortage of Increlex supply
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: W-TG-52800-010 (MS305)
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Primary Insulin-like Growth Factor-1 Deficiency
Keywords: Growth Hormone (GH) Insensitivity Syndrome; Insulin-like Growth Factor Deficiency (IGFD); Short Stature; Insulin-like Growth Factor (IGF-1); Growth
MeSH Terms: conditions — Dwarfism | interventions — mecasermin; Injections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Increlex patients: Eligible patients will be patients beginning therapy with Increlex® or those previously treated with Increlex.
  Interventions: Biological: mecasermin [rDNA origin] injection

INTERVENTIONS:
Biological: mecasermin [rDNA origin] injection — As prescribed by the physician.
  Other Names: Increlex®

SUMMARY:
This project is a retrospective (beginning January 2006) and prospective patient registry program sponsored by Ipsen (formerly Tercica, Inc.). In collaboration with participating health care practitioners, the patient registry program is an observational study monitoring the long-term safety of patients treated with Increlex® (mecasermin [rDNA origin] injection). The IGFD (Increlex® Growth Forum Database) Registry is intended primarily to monitor the safety and efficacy of Increlex replacement therapy in children with growth failure.

DETAILED DESCRIPTION:
The data collected for a patient will be those that exist in the patient's medical record as part of standard medical care. No additional patient procedures or activities are mandated by this study. The specific data to be collected at each visit and the schedule of data collection are listed in a schedule of assessments.

The collection of safety events is considered essential to the Registry. The website will provide the opportunity to report the occurrence of targeted adverse events (AEs), other important events considered to be related to Increlex administration and serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Parents or legally authorized representatives must give signed informed consent before any Registry-related activities are conducted. Assent from the subject should also be obtained where appropriate.
* Patients receiving Increlex® by a qualified practitioner may be enrolled

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be patients beginning therapy with Increlex® or those previously treated with Increlex.
Sampling Method: Non-Probability Sample
Enrollment: 1378 (Actual)
Dates: Start 2006-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To obtain long-term safety and efficacy data for Increlex® replacement therapy in children with growth failure | periodically assessed over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Endocrinology, Study Director — Ipsen (formerly Tercica)
Locations (1):
- Ipsen Central Contact, Basking Ridge, New Jersey, United States